CLINICAL TRIAL: NCT04722835
Title: Lung Macrophage Populations and Functions in Chronic Obstructive Pulmonary Disease (COPD)-Susceptible Smokers
Acronym: Pre-COPD Pilot
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of California, San Francisco (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 19-29768
Record Dates: First submitted 2020-12-09; First posted 2021-01-25 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Copd; Smoking; Tobacco Use
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking; Tobacco Use | interventions — Bronchoalveolar Lavage; Respiratory Physiological Phenomena; Blood Specimen Collection; Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 10 tablespoons of blood as well as Bronchoalveolar Lavage (BAL) samples will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal RV/TLC Group:: Plethysmographic RV/TLC equal or less than lower limit of normal.
  Interventions: Procedure: Bronchoscopy with Bronchoalveolar Lavage (BAL)
- Abnormal RV/TLC Group:: Plethysmographic RV/TLC higher than lower limit of normal.
  Interventions: Procedure: Bronchoscopy with Bronchoalveolar Lavage (BAL)

INTERVENTIONS:
Procedure: Bronchoscopy with Bronchoalveolar Lavage (BAL) — 1. Bronchoscopy w/ (BAL): The bronchoscope will be introduced through mouth and directed into the right middle lobe bronchus for bronchial lavage. The BAL will be performed with two 60-mL aliquots (total of 120 ml) of saline in each of medial and lateral segments of Right Middle Lobe (RML) (total 240 ml lavage).
  2. Albuterol Administration: The subjects will inhale 2 puffs of respiratory medication albuterol, then repeat the breathing test.
  3. Peak Flow Measurement: Subjects will breathe in fully then out forcefully into the handheld device.
  4. Pulmonary Function Test w/ Spirometry: will be used for determination of COPD and its severity. The PFT measures breathing capacity and lung function with different types of breathing maneuvers including flow-volume curve, single breath CO diffusing capacity, and total lung capacity.
  5. Blood draw
  6. Medical Health and Symptom Questionnaires
  7. Physical Exam by study doctor to determine suitability and safety for participation.
  Other Names: Albuterol Administration; Peak Flow Measurement; Pulmonary Function Test (with Spirometry); Blood draw; Medical Health and Symptom Questionnaires; Physical Exam

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a heterogeneous disease that affects only a fraction of those who smoke tobacco. The origin of this variability in susceptibility to develop COPD is unclear, but understanding its underlying biology has important implications for our ability to design suitable preventative and therapeutic strategies for its management. This Department of Defense (DOD) discovery research proposes to develop methodologies and generate preliminary data needed to lay the foundation for a large study that would investigate the underlying biological susceptibility of those who smoke tobacco to develop COPD.

DETAILED DESCRIPTION:
This is a pilot observational study of 20 subjects ≥40 years of age with smoking history of at least 20 pack-years (former or current) who have preserved spirometry, as defined by normal Forced Expiratory Volume (FEV1) / Forced Vital Capacity (FVC). Of the 20 subjects, 10 with and 10 without air trapping as determined by high and abnormal versus low and normal Residual Volume (RV) / Total Lung Capacity (TLC) measured by plethysmography. The cohort will undergo extensive clinical characterization including full Pulmonary Function Testing (PFT) and medical, symptom, activity, and quality of life questionnaires assessment including modified Medical Council Research (mMRC), COPD Assessment Test (CAT), Short Form-12 (SF12), and St. George's Respiratory (SGRQ) questionnaires. Subjects will undergo bronchoscopy with bronchoalveolar lavage (BAL) to obtain luminal macrophages and BAL fluid (BALF). Live BAL cells, BALF, and BAL cell RNA will be collected and stored in our biorepository for proposed studies. Molecular, functional, and transcriptomics analyses of luminal (alveolar) macrophages obtained by BAL (Aim 2) and protease activity measurement in serum and BALF will be performed (Aim 2) and will be examined against the clinical phenotype of the subjects, in particular air trapping-phenotype, to see if an underlying biological signature for susceptibility to develop COPD could be identified.

To perform a more comprehensive molecular and functional phenotype examination of lung macrophages, additional methodologies will be developed including a second mass cytometry (CyTOF) panel for single-cell proteomics and CyTOF-based phagocytosis and efferocytosis assays to allow for performance of truly single-cell functional phenotyping of myeloid cells from BAL and lung tissue (Aim 1).

ELIGIBILITY:
Inclusion Criteria:

* Ages between 40 to 75 years old.
* History of at least 20 pack-years of smoking.
* No diagnosis of COPD or asthma.
* No spirometric evidence of airflow obstruction as determined by FEV1/FVC ratio ≥0.7.
* FEV1 and FVC >lower limit of normal.
* Less than 1 pack-year history of tobacco smoking and no tobacco use within the past 12 months.
* Subjects will be divided into two groups by their RV/TLC:

Normal RV/TLC Group:

• Plethysmographic RV/TLC equal or less than lower limit of normal.

Abnormal RV/TLC Group:

• Plethysmographic RV/TLC higher than lower limit of normal.

Exclusion Criteria:

* Any history of IV drug use or inhalation of recreational drugs other than marijuana: A- within the past 20 years. B- more than 100 times IV drug usage. C- longer than 1 year usage.
* Marijuana use >400 joints in lifetime or any within past 6 months.
* Inability to walk briskly, run on treadmill, or pedal on ergometer to perform the study-required exercise level.
* Pregnant/breast feeding.
* Serious and active heart conditions- defined by stable or unstable angina, recent myocardial infarction (within the last 2 years), active congestive heart failure, ischemic cardiomyopathy.
* Liver cirrhosis.
* History of chronic active Hepatitis B or C.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The investigators will recruit both healthy, non-smoking subjects as well as subjects with at least 20 pack-years of smoking and air trapping.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of macrophage sub-populations in airway lumen. | 4 weeks
  Number of macrophages measured by flow cytometry.
Functional status of macrophage sub-populations in airway lumen. | 4 weeks
  Relative percentage of macrophages measured by flow cytometry.

SECONDARY OUTCOMES:
Symptomatic responses | 1 day
  Evidence for presence of mild exacerbation as measured by changes at or above the level of minimally clinically important difference (MCID) in each of the questionnaire's symptom score, 1-6, for the number of flare-ups in the past 3 years, with 6 being the worst outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Mehrdad Arjomandi, MD, Principal Investigator — University of California, San Francisco
Locations (3):
- United States (3):
  - Zuckerberg San Francisco General Hospital and Trauma Center, San Francisco, California
  - San Francisco VA Medical Center, San Francisco, California
  - University of California, San Francisco, San Francisco, California

IPD SHARING:
Plan to Share IPD: No